CLINICAL TRIAL: NCT04338503
Title: Mechanically Optimizing Cardiac Preload Using Partial Inferior Vena Cava Occlusion to Reduce Pulmonary Pressures in Heart Failure Patients in Heart Failure Patients
Brief Title: Mechanically Optimizing Cardiac Preload in Heart Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardioflow Technologies, LLC (Industry)
Collaborators: Saint Thomas Health (Other)
Responsible Party: Sponsor
Other Study IDs: CFT-37215-STH-01
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: pulmonary edema, preload
MeSH Terms: conditions — Heart Failure; Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HF patients: Decompensated heart failure patients undergoing right heart catheterization.
  Interventions: Diagnostic Test: Partial IVC occlusion

INTERVENTIONS:
Diagnostic Test: Partial IVC occlusion — Partial balloon occlusion of the inferior vena cava.

SUMMARY:
The purpose of the current study is to determine if partial balloon occlusion of the inferior vena cava can optimize cardiac pre-load and subsequently pulmonary pressures and cardiac output as a novel method to unload pulmonary edema and other symptoms of decompensated congestive heart failure. All products in this study are FDA approved and adhere to the specifications of the intended use.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled to undergo a right heart catheterization at Saint Thomas Hospital.
2. New York Heart Association (NYHA) II or III.
3. Subjects must be last least 18 years of age.
4. A left ventricular ejection fraction >= 20%.
5. Pulmonary artery occlusion pressure, or pulmonary wedge pressure >20 mmHg.

Exclusion Criteria:

1. Subjects without sinus rhythm.
2. Evidence of right heart failure.
3. Patients with primary pulmonary hypertension
4. Pulmonary wedge pressure <15mmHg.
5. Significant lung disease, such as prior diagnosis of COPD.
6. Resting or dynamic outflow tract gradient
7. Patients with left bundle branch block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Decompensated congestive heart failure patients referred for right heart catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary arterial pressures | During partial balloon occlusion
  Change in the measured mean pulmonary arterial pressure

SECONDARY OUTCOMES:
Change in cardiac output | During partial balloon occlusion
  Change in cardiac output measured in liters per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas Heart, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No